CLINICAL TRIAL: NCT05849285
Title: Evaluating a Model of Transitional and Lifelong Care for Adults With Childhood-Onset Disabilities
Brief Title: Evaluation of the Transitional and Lifelong Care Program
Status: Recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Laura Brunton, Assistant Professor, Western University, Canada
Other Study IDs: 122419; 184575 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2023-04-25; First posted 2023-05-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy; Spina Bifida; Developmental Disability
MeSH Terms: conditions — Cerebral Palsy; Spinal Dysraphism; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- TLC Patient: Patients of the TLC program with CP/SB/DD
  Interventions: Other: TLC Clinic
- Control Patient: Adults with CP/SB/DD that are not patients of the TLC Program
- TLC Caregiver: Caregiver of Patients of the TLC program with CP/SB/DD
  Interventions: Other: TLC Clinic
- Control Caregiver: Caregiver of Adults with CP/SB/DD that are not patients of the TLC Program
- Healthcare Providers: Healthcare Providers who care for patients in the TLC clinic
  Interventions: Other: TLC Clinic

INTERVENTIONS:
Other: TLC Clinic — Patients of the TLC clinic - receive coordinated multidisciplinary and specialized care from a team
  Groups: Healthcare Providers; TLC Caregiver; TLC Patient

SUMMARY:
The population cared for in the Transitional and Lifelong Care (TLC) clinic is youth and adults with childhood-onset disability, of which the large majority are adults with brain-based, neurodevelopmental conditions such as cerebral palsy, spina bifida and developmental disability. The TLC program was created to address the health inequities that have long existed for this population because of the gaps in care they experience once they transition from pediatric healthcare services to the adult healthcare sector. The TLC program offers coordinated and comprehensive management of co-occurring mental, social and physical health conditions for this group of adults with neurodiverse conditions. The proposed study will provide much needed evaluation of the TLC model as an intervention to provide transitional and lifelong care that reduces the barriers experienced because of the undefined clinic path - potentially more appropriately referred to as a "cliff" by a Freeman et al., (2015) - for these individuals. With appropriate evidence of effectiveness, scaling of the TLC program to other Ontario Health regions and more widely across Canada would improve access healthcare providers who are knowledgeable and competent in the management of physical and mental health conditions for adults with neurodiverse conditions as well as service integration and coordination between social and health sectors. The TLC clinic was co-designed with adults with neurodiverse conditions and health care providers in 2014 and represents a significant and sustainable change in the way healthcare has been delivered for this population in the Ontario Health West region over the last 7 years. More than 750 people have accessed coordinated and comprehensive care from Physiatrists, a Nurse Practitioner, Social Worker, Physiotherapist, Occupational Therapist, Speech Language Pathologist, Registered Dietitian and Rehabilitation Therapist in the TLC program since it began, documenting the effectiveness of this care has the power to re-shape care received for adults with neurodiverse conditions that onset in childhood in Canada.

ELIGIBILITY:
Inclusion Criteria:

Each participant dyad will consist of one person, of either sex and gender, who is over the age of 21 years with a childhood-onset disability, and the primary caregiver (based on contact hours) or support person, of either sex and gender, involved in their care. In cases where the patient participant is independent with care, a spouse or family member may still participate in the caregiver portion of the study.

2. Patient participants will have continuously resided in Ontario during the years of 2015 to 2020 to facilitate full data retrieval from the administrative dataset.

3. Healthcare providers, of any discipline, who provide care to adults with childhood-onset conditions in the TLC program.

Exclusion Criteria:

Patient participants will be ineligible if they are in a phase of deterioration associated with a progressive health condition identified either personally or by the caregiver participant.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be categorized into two cohorts: 1) patients of the TLC program, 2) controls . Participant dyads will be formed that include the adult patient (and a caregiver, spouse, or support person that may be involved in the patient's care. TLC dyads will be recruited from the existing client base of the program and control dyads will be recruited from the Kitchener/Waterloo/Cambridge area of Ontario (and the surrounding rural areas).
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | Year 1
  MPOC-A (Measure of Processes of Care - Adults) Each domain score, ranging from 0.0 to 7.0, is computed by averaging the ratings for the items of that domain, higher scores represent better outcomes

SECONDARY OUTCOMES:
Health Related Quality of Life (General) | Year 1
  EQ5D5L The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression). The descriptive system describes 3125 (=5⁵) potential health states.
Health Related Quality of Life (WHO) | Year 1
  WHOQOL-BREF (World Health Organization Quality of Life - Brief) Lowest and highest possible scores to zero and 100, respectively. Higher scores represent better outcomes
Caregiver Burden | Year 1
  BSFC (Burden Scale for Family Caregivers). Minimum score is 0, maximum score is 84, higher scores represent worse outcome (more burden).
Perceived Support of Healthcare Providers | Year 1
  MPOC-SP (Measure of Processes of Care - Service Providers). Each domain score, ranging from 0.0 to 7.0, is computed by averaging the ratings for the items of that domain, higher scores represent better outcomes
Economic Analysis | Year 2
  Unit Costs of healthcare used

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Brunton, PhD, Principal Investigator — Western University
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be available to share upon request made by other researchers once a plan of analysis has been proposed to the team